CLINICAL TRIAL: NCT00485433
Title: A Phase 2 Multicenter, Randomized, Double-blind, Parallel-group, Active-control, Dose-ranging Study to Evaluate the Safety and Efficacy of a Single Administration of SKY0402 for Prolonged Postoperative Analgesia in Subjects Undergoing Primary Unilateral Inguinal Hernia Repair.
Brief Title: Dose-ranging Study for Postoperative Analgesia in Subjects Undergoing Primary Unilateral Inguinal Hernia Repair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SKY0402-C-207
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain
Keywords: hernia; unilateral; postoperative; analgesia
MeSH Terms: conditions — Pain, Postoperative; Hernia; Agnosia | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bupivacaine HCl 105mg (Active Comparator): Bupivacaine HCl given during hernia repair
  Interventions: Drug: Bupivacaine HCl
- SKY0402 low dose (Experimental): SKY0402 low dose given during hernia repair
  Interventions: Drug: SKY0402
- SKY0402 Middle dose (Experimental): SKY0402 middle dose given during hernia repair
  Interventions: Drug: SKY0402
- SKY0402 High dose (Experimental): SKY0402 high dose given during hernia repair
  Interventions: Drug: SKY0402

INTERVENTIONS:
Drug: Bupivacaine HCl — Bupivacaine HCl given during hernia repair
  Other Names: Marcaine 0.25% with epinephrine 1:200,000
  Arms: Bupivacaine HCl 105mg
Drug: SKY0402 — SKY0402 given during hernia repair
  Other Names: EXPAREL
  Arms: SKY0402 High dose; SKY0402 Middle dose; SKY0402 low dose

SUMMARY:
The purpose of this study is to evaluate three dose levels of SKY0402 compared with 105 mg of bupivacaine HCl.

DETAILED DESCRIPTION:
Effective postoperative pain control is a critical element in patient recovery, as the majority of patients may experience significant pain, particularly in the first few days following surgery. Appropriate postoperative pain management contributes to improved healing, faster patient mobilization, shortened hospital stays, and reduced healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. Males 18 years of age and older at the Screening Visit.
2. Scheduled to undergo, elective, primary, unilateral, open-technique, tension-free (Lichtenstein-type technique with mesh) inguinal hernia repair under general anesthesia.
3. American Society of Anesthesiology (ASA) Physical Class 1-3.
4. Capable and willing to comply with all study visits and procedures and to provide written informed consent.
5. Able to speak, read, and understand the language of the informed consent form, study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments.

Exclusion Criteria:

1. Use of any of the following medications within the times specified before surgery:

   * Long-acting opioid medication within 3 days.
   * Any opioid medication within 24 hours.
2. Concurrent painful physical condition that may require analgesic treatment in the postoperative period for pain that is not strictly related to the hernia repair procedure and may confound the postoperative assessments (e.g., rheumatoid arthritis, neuropathic pain, concomitant vasectomy).
3. Body weight less than 50 kilograms.
4. History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics.
5. Other contraindication to bupivacaine.
6. Contraindication(s) to epinephrine, such as concurrent administration of monoamine oxidase (MAO) inhibitors or antidepressants of amitriptyline or imipramine types, conditions where the production or exacerbation of tachycardia could prove fatal (e.g., poorly controlled thyrotoxicosis or severe heart disease), or any other pathological conditions that might be aggravated by the effects of epinephrine.
7. Contraindication to any of the pain control agents anticipated to be used postoperatively (i.e., acetaminophen or oxycodone).
8. Administration of an investigational product within 30 days or 5 elimination half-lives of such investigational product, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
9. Suspected or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
10. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.
11. Current or historical evidence of any clinically significant condition that, in the opinion of the Investigator, may increase the risk of surgery, complicate the subject's postoperative course, or indicate an increased vulnerability to study drugs and procedures and expose the subject to an unreasonable risk as a result of participating in this clinical trial.

    If during surgery the following criterion is met:
12. Any clinically significant event or condition uncovered during the hernia repair surgery (e.g., excessive bleeding) that might render the subject medically unstable or complicate the subject's postoperative course.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arcadia Methodist Hospital, Arcadia, California
  - Saddleback Valley Outpatient Surgery, Laguna Hills, California
  - Huntington Memorial Hospital, Pasadena, California
  - St. Luke's Roosevelt Hosptial Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Memorial Hermann Healthcare System, Houston, Texas
  - Kirby Outpatient Surgical Center, Houston, Texas

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine HCl 105mg | SKY0402 Low Dose | SKY0402 Middle Dose | SKY0402 High Dose
Started | 24 | 25 | 24 | 25
Completed | 24 | 25 | 24 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine HCl 105mg | SKY0402 Low Dose | SKY0402 Middle Dose | SKY0402 High Dose | Total
Number analyzed (Participants) | 24 | 25 | 24 | 25 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 18 | 21 | 79
  >=65 years | 3 | 6 | 6 | 4 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (16.9) | 51.2 (17.3) | 54 (15.1) | 52.1 (15.6) | 51.1 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 24 | 25 | 24 | 25 | 98
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 24 | 25 | 98

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) With Activity (NRS-A) Pain Intensity Scores From 0 Through 72 Hours
Description: The subject's pain intensity was to be assessed with activity (NRS-A), after the subject had moved himself from a supine position in bed to a sitting up position at the edge of the bed. The subject was to respond to the following question: "On a scale of 0 to 10, where 0=no pain and 10=worst possible pain, how much pain did you have while sitting up?"
Time Frame: 0 to 72 hours
Measure: Mean (Standard Deviation); unit: Units on a scale*hours
Groups:
- Bupivacaine HCl 105mg: A single dose of 105 mg bupivacaine in a 42-mL injection volume administered via local infiltration during surgery
- SKY0402 Low Dose: A single dose of SKY0402 105mg diluted to a 42-mL injection volume administered via local infiltration during surgery
- SKY0402 Middle Dose: A single dose of SKY0402 180mg diluted to a 42-mL injection volume administered via local infiltration during surgery
- SKY0402 High Dose: A single dose of SKY0402 345 mg diluted to a 42-mL injection volume administered via local infiltration during surgery
Arm/Group | Bupivacaine HCl 105mg | SKY0402 Low Dose | SKY0402 Middle Dose | SKY0402 High Dose
Number analyzed (Participants) | 24 | 25 | 24 | 25
Units on a scale*hours | 298.1 (136.6) | 286.9 (146.4) | 274.6 (115.4) | 274.4 (253.4)

2. Secondary Outcome: Number of Participants With Adverse Events Through 96 Hours or Serious Adverse Events Through 30 Days
Time Frame: Up to 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- SKY0402 (All Doses): SKY0402 given during hernia repair
Arm/Group | Bupivacaine HCl 105mg | SKY0402 (All Doses)
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/74
Other Adverse Events (participants affected / at risk) | 10/24 | 17/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine HCl 105mg (N=24) | SKY0402 (All Doses) (N=74)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Occurred in the Low Dose group
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine HCl 105mg (N=24) | SKY0402 (All Doses) (N=74)
Nausea (Gastrointestinal disorders) | 5 | 6
Constipation (Gastrointestinal disorders) | 2 | 7
Dizziness (Nervous system disorders) | 2 | 6
Hypoaesthesia (Nervous system disorders) | 2 | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No